CLINICAL TRIAL: NCT06522698
Title: Optimizing Research Data Acquisition With Smart Pill Bottles: A Feasibility and Implementation Study
Brief Title: Optimizing Research Data Acquisition With Smart Pill Bottles
Acronym: SPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Pascal Laferrière-Langlois, Clinical assistant professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-3801
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain; Opioid Use
Keywords: Major abdominal surgery; Connected Technology; Chronic Pain; Postoperative pain; Opioid consumption; Smart Pill Bottles
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smart Pill Bottle Data Collection Group (Experimental): Group of patients in which data on postoperative opioid medication consumption will be collected through the use of smart pill bottles.
  Interventions: Device: Smart Pill Bottle

INTERVENTIONS:
Device: Smart Pill Bottle — Patients in the intervention group will have their opioid medication consumption monitored through a smart pill bottle that records medication usage and streamlines the data into an online platform accessible by the medical staff. This group will also fill out surveys delivered through the smart pill bottle's online platform.
  Other Names: Connected Pill Bottle

SUMMARY:
The goal of this clinical trial is to learn if smart pill bottles can be used as a tool to optimize data collection in clinical trials by increasing the quality of data collected and limiting the associated cost. The main questions it aims to answer are:

Is the use of smart pill bottles a feasible method of data collection in clinical trials in terms of patient adherence.

Is the data collected by the smart pill bottles of higher quality than that collected through human resources? What is the impact of the use of smart pill bottles on the costs involved in clinical trials ?

Researchers will collect data on postoperative opioid medication consumption with the smart pill bottle and assess the adherence of patients to the device along with the quality of data collected and the costs involved in the process.

Participants will:

Use the smart pill bottle to consume opioid medication following surgery for 3 months At the end of the 3 month period, the group will have filled out surveys detailing their opioid consumption, surgical pain and other relevant information.

DETAILED DESCRIPTION:
Several studies involving harnessing new technology to approach data collection have suggested that a streamlined and automated method of collecting data through connected technology can help set up cohort studies more cost-effectively. Evaluating the use of a connected device as a research tool in clinical trials and comparing it with traditional data collection using human resources would provide valuable insights into its efficiency and effectiveness. Smart medication adherence monitoring devices are a novel technology that provides objective and granular medication utilization data along with engaging patients with their treatment. Particularly, the smart pill bottle (SPB) is a rapidly developing technology that allows for medication monitoring of solid doses with the use of electronic sensors that can collect data on medication usage in real time and offer direct communication between patients and healthcare professionals or trialists. SPBs have shown efficacy in monitoring compliance and possibly increasing medication adherence in the clinical setting and the technology has been suggested as a potential research tool that would allow automatic collection of granular and precise data on the time of medication intake, dose, and frequency. However, there hasn't been a trial comparing the efficacy of using SPBs for data collection in clinical trials versus the traditional method reliant on human resources in comparable contexts. Based on the properties of SPBs and available literature supporting the automatization and streamlining of data in clinical trials, the investigators believe that the use of these devices may allow data collection of higher quality regarding granularity, number of losses of follow-up, completeness, missing data points along with a reduction of costs incurred by avoiding the use of human resources.

The aim of this study is to evaluate the feasibility of using smart pill bottles (SPBs) to optimize data collection in the context of randomized control trials.

The project will be a prospective observational study conducted at the CIUSSS-de-l'Est-de-l'Île-de-Montréal (Hôpital Maisonneuve-Rosemont) over a period of 6 to 12 months.

To do so, 155 patients undergoing major abdominal surgery with postoperative opioid medication prescription will be recruited. These patient's medication consumption will be monitored with the use of a smart pill bottle for a duration of 90 days. The results of this cohort will be compared with a historical cohort from a previous study conducted within the same hospital network. The protocol for the current trial was purposefully designed to be comparable to that of this historical cohort.

A loan of 50 SPBs will be obtained from Thess Corporate (Company producing smart pill bottles).

ELIGIBILITY:
Inclusion Criteria:

* All consenting adult patients (age >17 years) undergoing major abdominal surgery via laparotomy (any open surgery involving the abdominal compartment or its wall, excluding appendectomies, inguinal hernia repairs, abdominal wall hernia repairs, and incisional hernia repairs)

Exclusion Criteria:

* Patients enrolled in the historical cohort (POCAS study)
* Patients currently participating in another study
* Patients planned to undergo additional surgery within 90 days after the surgery
* Patients who do not understand French or English.
* Patients planned to be redirected to a secondary care or rehabilitation establishment following discharge
* Patients with diagnosed cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to data collection method | 3 months
  The percentage of patients that will have used the smart pill bottle (SPB) until the end of the 90-day period or until the absence of pain, as opposed to any change in medication intake strategy that results in ceasing the use of the SPB. (High percentage is a better outcome)

SECONDARY OUTCOMES:
The quality of data acquired through the SPBs | 3 months
  The granularity of data acquired, the preciseness of data points, the number of loss of follow-up compared with the historical cohort from the POCAS study which collected data from a comparable patient group through human resources.
The costs incurred from carrying out the project | 3 months
  The costs incurred from carrying out the project compared with the historical cohort from the POCAS study which collected data from a comparable patient group through human resources.
The time for recruitment of patients | Up to12 months
  The time for recruitment of patients compared with the historical cohort from the POCAS study which collected data from a comparable patient group through human resources. (Lower time is a better outcome)
Prevalence of persistent opioid consumption 90 days after surgery | 7 days
  Persistent opioid consumption (POC) 90 days after surgery as reported by the SPBs. POC will be defined as consumption of any quantity of opioids in the 7 days prior to the 90-day interrogation. This definition will be accurate for both preoperative chronic and non-chronic opioid users. (Higher rate of persistent consumption is a worse outcome)
Prevalence of Chronic post-surgical pain 90 days after surgery | 7 days
  The presence of chronic post-surgical pain (CPSP) in the 7 days prior to the interrogation (interrogation occurs at 90 days post-op). CPSP will be defined as any pain at the surgical site for patients who had pain at that site before surgery (by 1 point on the general numerical pain scoring question of the BPI questionnaire) (12).
Change in Quality of Life | 3 months
  The change in the reported quality of life at 90 days post-op. QOL will be measured as a continuous variable on the SF-12 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laferriere-Langlois, MD, MSc, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catala-Lopez F, Aleixandre-Benavent R, Caulley L, Hutton B, Tabares-Seisdedos R, Moher D, Alonso-Arroyo A. Global mapping of randomised trials related articles published in high-impact-factor medical journals: a cross-sectional analysis. Trials. 2020 Jan 7;21(1):34. doi: 10.1186/s13063-019-3944-9. PMID 31910857
- [Background] Vinkers CH, Lamberink HJ, Tijdink JK, Heus P, Bouter L, Glasziou P, Moher D, Damen JA, Hooft L, Otte WM. The methodological quality of 176,620 randomized controlled trials published between 1966 and 2018 reveals a positive trend but also an urgent need for improvement. PLoS Biol. 2021 Apr 19;19(4):e3001162. doi: 10.1371/journal.pbio.3001162. eCollection 2021 Apr. PMID 33872298
- [Background] Setia MS. Methodology Series Module 1: Cohort Studies. Indian J Dermatol. 2016 Jan-Feb;61(1):21-5. doi: 10.4103/0019-5154.174011. PMID 26955090
- [Background] Toledano MB, Smith RB, Brook JP, Douglass M, Elliott P. How to Establish and Follow up a Large Prospective Cohort Study in the 21st Century--Lessons from UK COSMOS. PLoS One. 2015 Jul 6;10(7):e0131521. doi: 10.1371/journal.pone.0131521. eCollection 2015. PMID 26147611
- [Background] Barrera-Valencia C, Perea-Florez EX. Comparison of Costs in Teledermatology Using PC and Camera Versus Smartphone. Telemed J E Health. 2024 Jun;30(7):e2087-e2095. doi: 10.1089/tmj.2023.0369. Epub 2024 Apr 26. PMID 38669106
- [Background] Pavlovic I, Miklavcic D. Web-based electronic data collection system to support electrochemotherapy clinical trial. IEEE Trans Inf Technol Biomed. 2007 Mar;11(2):222-30. doi: 10.1109/titb.2006.879581. PMID 17390992
- [Background] Zijp TR, Touw DJ, van Boven JFM. User Acceptability and Technical Robustness Evaluation of a Novel Smart Pill Bottle Prototype Designed to Support Medication Adherence. Patient Prefer Adherence. 2020 Mar 20;14:625-634. doi: 10.2147/PPA.S240443. eCollection 2020. PMID 32256053
- [Background] Aldeer M, Javanmard M, Martin RP. A Review of Medication Adherence Monitoring Technologies. Applied System Innovation. 2018; 1(2):14. https://doi.org/10.3390/asi1020014
- [Background] Schwed A, Fallab CL, Burnier M, Waeber B, Kappenberger L, Burnand B, Darioli R. Electronic monitoring of compliance to lipid-lowering therapy in clinical practice. J Clin Pharmacol. 1999 Apr;39(4):402-9. doi: 10.1177/00912709922007976. PMID 10197299
- [Background] Ellsworth GB, Burke LA, Wells MT, Mishra S, Caffrey M, Liddle D, Madhava M, O'Neal C, Anderson PL, Bushman L, Ellison L, Stein J, Gulick RM. Randomized Pilot Study of an Advanced Smart-Pill Bottle as an Adherence Intervention in Patients With HIV on Antiretroviral Treatment. J Acquir Immune Defic Syndr. 2021 Jan 1;86(1):73-80. doi: 10.1097/QAI.0000000000002519. PMID 33306564
- [Background] Toscos T, Drouin M, Pater JA, Flanagan M, Wagner S, Coupe A, Ahmed R, Mirro MJ. Medication adherence for atrial fibrillation patients: triangulating measures from a smart pill bottle, e-prescribing software, and patient communication through the electronic health record. JAMIA Open. 2020 Apr 28;3(2):233-242. doi: 10.1093/jamiaopen/ooaa007. eCollection 2020 Jul. PMID 32734164
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Huo T, Guo Y, Shenkman E, Muller K. Assessing the reliability of the short form 12 (SF-12) health survey in adults with mental health conditions: a report from the wellness incentive and navigation (WIN) study. Health Qual Life Outcomes. 2018 Feb 13;16(1):34. doi: 10.1186/s12955-018-0858-2. PMID 29439718
- [Background] Nafziger AN, Barkin RL. Opioid Therapy in Acute and Chronic Pain. J Clin Pharmacol. 2018 Sep;58(9):1111-1122. doi: 10.1002/jcph.1276. Epub 2018 Jul 9. PMID 29985526
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Page MG, Kudrina I, Zomahoun HTV, Croteau J, Ziegler D, Ngangue P, Martin E, Fortier M, Boisvert EE, Beaulieu P, Charbonneau C, Cogan J, Daoust R, Martel MO, Neron A, Richebe P, Clarke H. A Systematic Review of the Relative Frequency and Risk Factors for Prolonged Opioid Prescription Following Surgery and Trauma Among Adults. Ann Surg. 2020 May;271(5):845-854. doi: 10.1097/SLA.0000000000003403. No abstract available. PMID 31188226
- [Background] https://www.thess-corp.fr/
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Schirle L, Stone AL, Morris MC, Osmundson SS, Walker PD, Dietrich MS, Bruehl S. Leftover opioids following adult surgical procedures: a systematic review and meta-analysis. Syst Rev. 2020 Jun 11;9(1):139. doi: 10.1186/s13643-020-01393-8. PMID 32527307